CLINICAL TRIAL: NCT06620874
Title: Comparison of the Efficacy of Ultrasound-Guided Injections of Saline, High-Concentration Dextrose, and Ligament Repair Agents for the Treatment of Medial Collateral Ligament Pathology in Degenerative Knee Osteoarthritis: A Randomized Double-Blind Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Ting-an (Other)
Responsible Party: Sponsor-Investigator, Chen Ting-an, Attending Physician, Shin Kong Wu Ho-Su Memorial Hospital
Organization: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20240724R
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Medial Collateral Ligament Lesions; Knee Osteoarthritis
Keywords: medical collateral ligament (MCL); Knee osteoarthritis; prolotherapy; STABHA; rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STABHA Injection (Experimental): Participants will receive two ultrasound-guided STABHA injections into the medial collateral ligament of the knee at a 2-week interval.
  Interventions: Biological: STABHA Injection
- High-Concentration Glucose Water Injection (Experimental): Participants will receive two ultrasound-guided high-concentration glucose water injections into the medial collateral ligament of the knee at a 2-week interval.
  Interventions: Other: High-Concentration Glucose Water Injection
- Saline Injection (Placebo Comparator): Participants will receive two ultrasound-guided saline injections into the medial collateral ligament of the knee at a 2-week interval.
  Interventions: Other: Saline Injection

INTERVENTIONS:
Biological: STABHA Injection — Participants will receive two ultrasound-guided STABHA injections into the medial collateral ligament of the knee at a 2-week interval
  Arms: STABHA Injection
Other: High-Concentration Glucose Water Injection — Participants will receive two ultrasound-guided high-concentration glucose water injections into the medial collateral ligament of the knee at a 2-week interval
  Arms: High-Concentration Glucose Water Injection
Other: Saline Injection — Participants will receive two ultrasound-guided saline injections into the medial collateral ligament of the knee at a 2-week interval
  Arms: Saline Injection

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of STABHA, high-concentration glucose water, and saline injections in treating knee osteoarthritis with medial collateral ligament lesions. This prospective, double-blind, randomized trial will recruit 51 patients from the Shin Kong Hospital Rehabilitation Department.

The main questions it aims to answer are:

1. Do STABHA or high-concentration glucose water injections provide better pain relief and improved knee function compared to saline?
2. What side effects do participants experience with these treatments?

Participants will be randomly divided into three groups: STABHA, high-concentration glucose water, and saline. In addition to routine intra-articular hyaluronic acid injections, each group will receive two ultrasound-guided injections of their assigned treatment into the medial collateral ligament of the knee, with a two-week interval. All participants will also undergo a 4-week physical therapy program.

Participants will:

1. Receive two ultrasound-guided injections over two weeks.
2. Undergo 4 weeks of physical therapy.
3. Return for follow-up assessments at 1 and 3 months, including the WOMAC osteoarthritis index, pain score, KOOS knee outcome score, knee range of motion, and knee ultrasound examination.

ELIGIBILITY:
Inclusion Criteria:

-

The patients should fulfill the following criteria:

1. Age between 45 to 80 years old.
2. Meet at least three of the six American College of Rheumatology (ACR) criteria, including age over 50 years, morning stiffness less than 30 minutes, crepitus in passive knee movements, bony tenderness, bony enlargement, and no palpable warmth.
3. Radiologic grading of 2 or 3 according to Kellgren-Lawrence criteria.
4. Evidence of medial collateral ligament (MCL) pathology with incomplete injuries (grade I or II).
5. Willing to receive prolotherapy treatment.
6. Willing and able to complete all follow-ups and assessments in the randomized double-blind trial.

Exclusion Criteria:

* The exclusion criteria are:

  1. Severe systemic disorders including cancer, uncontrolled diabetes mellitus, sepsis, or cardiopulmonary diseases.
  2. History of anticoagulation therapy, knee injection over the past three months.
  3. History of knee surgery or candidates for knee arthroplasty.
  4. History of intolerance to prolotherapy.
  5. Pregnancy.
  6. Infectious arthritis, inflammatory joint diseases, joint dysplasia.
  7. Body Mass Index (BMI) greater than 35 kg/m2.
  8. Complete tear of medial collateral ligament under ultrasound.
  9. Fracture or other causes of knee pain instead of osteoarthritis.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction Using WOMAC Osteoarthritis Index | Baseline, 1 month, and 3 months post-intervention
  The primary outcome will assess the change in pain scores using the WOMAC Osteoarthritis Index at baseline, 1 month, and 3 months after the treatment intervention

SECONDARY OUTCOMES:
Knee Range of Motion | Baseline, 1 month, and 3 months post-intervention
  The change in knee range of motion will be measured using a goniometer at baseline, 1 month, and 3 months after intervention
KOOS Knee Outcome Score | Baseline, 1 month, and 3 months post-intervention
  The outcome will assess the change in KOOS Knee Outcome Score at baseline, 1 month, and 3 months after the treatment intervention

OTHER OUTCOMES:
Change in Medial Collateral Ligament (MCL) Characteristics in Knee Ultrasound Examination | Baseline, 1 month, and 3 months post-intervention
  The outcome will assess changes in the characteristics of the medial collateral ligament (MCL) of the knee using ultrasound examination. Measurements will include MCL thickness, echogenicity, and presence of any structural abnormalities (e.g., calcifications, tears). Ultrasound evaluations will be performed at baseline, 1 month, and 3 months after the intervention to determine the treatment effects on MCL condition.

IPD SHARING:
Plan to Share IPD: No